CLINICAL TRIAL: NCT04832789
Title: Ultra-Low Tidal Volume Mechanical Ventilation in ARDS Through ECMO (ULTIMATE) Pilot Randomized Trial
Brief Title: Ultra-Low Tidal Volume Mechanical Ventilation in ARDS Through ECMO
Acronym: ULTIMATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Eddy Fan, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ULTIMATE
Record Dates: First submitted 2021-03-28; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: ARDS
Keywords: ECMO; Mechanical Ventilation; Ventilator-induced lung injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Best conventional ventilation (No Intervention)
- Ultra-protective ventilation with ECMO (Experimental)
  Interventions: Device: Venovenous ECMO

INTERVENTIONS:
Device: Venovenous ECMO — Venovenous ECMO
  Arms: Ultra-protective ventilation with ECMO

SUMMARY:
Primary Research Question for the Full ULTIMATE Randomized Clinical Trial (RCT): What is the effect of ultra-protective ventilation facilitated by extracorporeal membrane oxygenation (ECMO) versus best current conventional ventilation (CV) on all-cause hospital mortality among patients with early moderate-severe acute respiratory distress syndrome (ARDS)?

Secondary Research Questions: Among patients with early moderate-severe ARDS, what is the effect of ultra-protective ventilation versus CV on: (1) duration of mechanical ventilation; (2) duration of ICU and hospital stay; (3) organ dysfunction; (4) barotrauma; and (5) mortality at other time-points (ICU discharge, 28-day, 60-day)?

The ULTIMATE Pilot Study: Before embarking on a definitive multinational trial to address the questions listed above, the ULTIMATE Pilot Study has these 3 specific feasibility objectives:

1. To assess adherence to our explicit mechanical ventilation protocols, with particular focus on delivered tidal volumes in both groups;
2. To estimate the rate of patient recruitment and understand barriers to recruitment; and
3. To measure and understand the reasons for crossovers or rescue by ECMO in the control group.

In addition, we will monitor safety issues, recording serious adverse events in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Endotracheal mechanical ventilation for ≤ 5 days
3. Early moderate-severe ARDS (Berlin Definition) - all of the following conditions for ≤ 48 hours i. PaO2/FiO2 ≤200 with PEEP > 5 cmH2O ii. bilateral opacities not fully explained by effusions, lobar/lung collapse, or nodules iii. respiratory failure not fully explained by cardiac failure or fluid overload iv. within one week of a known insult of new or worsening respiratory symptoms
4. ARDS severity criterion - either 1 of:

   1. PaO2/FiO2 ≤ 150 mm Hg, on PEEP ≥ 10 cm H2O and FiO2 ≥ 0.5

Exclusion Criteria:

1. Currently receiving any form of ECMO (e.g., venovenous, venoarterial, or hybrid configuration)
2. Chronic hypercapnic respiratory failure defined as PaCO2 > 60 mmHg in the outpatient setting
3. Home mechanical ventilation (non-invasive ventilation or via tracheotomy), not CPAP
4. Actual body weight exceeding 1 kg per centimeter of height
5. Severe hypoxemia with PaO2/FiO2 < 80 mmHg
6. Expected mechanical ventilation duration < 48 hours
7. Treating team is in the process of moving to a palliative mode of care
8. Moribund patient not expected to survive 24 hours despite ongoing life-sustaining therapies
9. Confirmed diffuse alveolar hemorrhage from vasculitis
10. Contraindications to limited anticoagulation (e.g., active GI bleeding, bleeding diathesis)
11. Pregnancy - due to unknown effects of PaCO2 changes on placental blood flow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients adhering to the study protocol | Through study completion, an average of 2 years
  Adherence to our explicit ventilation protocols will be adequate if more than 80% of patients have fewer than 10% of monitored values as major protocol violations
Proportion of patients crossing over to VV ECMO | Through study completion, an average of 2 years
  The number of protocol withdrawals or off-protocol treatment with VV ECMO will be acceptable if fewer than 10% of patients crossover or receive VV ECMO, when not allowed by the protocol
Number of patients recruited for the study | Through study completion, an average of 2 years
  Patient accrual will be adequate if we recruit 72 patients from 12 sites over 1 year of enrolment

SECONDARY OUTCOMES:
Ventilator-free days | Up to 30 days
  Duration of alive and free of invasive mechanical ventilation
Length of stay | Through study completion, an average of 2 years
  ICU and hospital length of stay in survivors and non-survivors
Number of patients with non-pulmonary organ dysfunction | Up to 30 days
  Using standard definitions
Number of patients with barotrauma | Up to 30 days
  New barotrauma
Mortality | Through study completion, an average of 2 years
  At ICU discharge and 30-days
Health-related quality of life | At 6 months post-randomization
  Health-related quality of life (EQ-5D) via telephone

CONTACTS AND LOCATIONS:
Overall Officials: Niall Ferguson, MD, MSc, Principal Investigator — University Health Network, Toronto; Eddy Fan, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (11):
- United States (2):
  - New York Presbyterian Hospital, New York, New York
  - OHSU Hospital, Portland, Oregon
- Canada (9):
  - University of Alberta Hospital, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Unity Health, Toronto, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec